CLINICAL TRIAL: NCT03277001
Title: Multi-center、Randomize、Open、Non-inferiority Study of Prophylactic Effect of Rivaroxaban on Venous Thromboembolism in AECOPD
Brief Title: Study of Prophylactic Effect of Rivaroxaban on Venous Thromboembolism in AECOPD
Acronym: SUPREME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Shengqing Li, Chief physician, Professor-levelled doctor, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2017-279
Record Dates: First submitted 2017-09-02; First posted 2017-09-08 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Acute Exacerbation Copd; Venous Thromboembolism
Keywords: AECOPD; VTE prevention; Rivaroxaban; LMWHs
MeSH Terms: conditions — Venous Thromboembolism | interventions — Rivaroxaban; Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enoxaparin (Active Comparator): AECOPD patients meeting the eligibility criterion by GOLD2017 in hospitalization Padua score > 4
  Interventions: Drug: Enoxaparin
- Rivaroxaban (Experimental): AECOPD patients meeting the eligibility criterion by GOLD2017 in hospitalization Padua score > 4
  Interventions: Drug: Rivaroxaban

INTERVENTIONS:
Drug: Rivaroxaban — Rivaroxaban, po. 10mg/day（CrCl≥ 50 ml/min）or 5 mg /day (CrCl ≥ 30 and < 50 ml/min) po.
  Arms: Rivaroxaban
Drug: Enoxaparin — Enoxaparin 40mg IH
  Arms: Enoxaparin

SUMMARY:
AECOPD increases the risk of VTE.VTE prevention is a long way to go for high-risk VTE patients in China.The incidence of AECOPD complicated with VTE in Asian population is high and the mortality rate is high.Rivaroxaban, a new oral anticoagulant, has been widely used in the treatment and prevention of VTE.However the question about the efficacy and safety of new oral anticoagulant compared with LMWHs for the prevention of symptomatic VTE and VTE-related death post-hospital discharge in high-risk AECOPD patients is still unknown. Thus this study is to evaluate if the prophylactic anticoagulation effect by Rivaroxaban is non-inferiority than Enoxaprine in high risk AECOPD and to evaluate the safety of using Rivaroxaban to prevent VTE in high risk AECOPD comparing with Enoxaprine.

DETAILED DESCRIPTION:
The acute exacerbation of COPD increases the risk of venous thromboembolism.VTE prevention is a long way to go for high-risk VTE patients in China.The incidence of AECOPD complicated with VTE in Asian population is high and the mortality rate is high.Rivaroxaban, a new oral anticoagulant, has been widely used in the treatment and prevention of VTE.However the question about the efficacy and safety of new oral anticoagulant compared with LMWHs for the prevention of symptomatic VTE and VTE-related death post-hospital discharge in high-risk AECOPD patients is still unknown. Thus this study is to evaluate if the prophylactic anticoagulation effect by Rivaroxaban is non-inferiority than Enoxaprine in high risk AECOPD and to evaluate the safety of using Rivaroxaban to prevent VTE in high risk AECOPD comparing with Enoxaprine.

ELIGIBILITY:
Inclusion Criteria:

* AECOPD patients meeting the eligibility criterion by GOLD2017 in hospitalization；Padua score > 4；Age from 40-80y

Exclusion Criteria:

* Patients whose admitting diagnosis was VTE；Patients whose duration of hospital stay was <3 days or >30 days ；Patients who received therapeutic doses of anticoagulants or thrombolytic therapy for any indication before hospitalization；an organic lesion that could bleed; severe liver or renal failure; confirmed or uncontrolled hypertension; a congenital or acquired coagulation disorder; a history of hypersensitivity or thrombocytopenia to heparins of any type；Patients who were contraindicated to anticoagulant therapy, venography, or angiography

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 438 (Estimated)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2019-07-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
VTE incidence | 1 month
  VTE incidence ( include PE and DVT)

SECONDARY OUTCOMES:
In-hospital Motality | 1 month
  in-hospital Motality
Hospital duration | 1 month
  length of hospital stay
incidence of bleeding | 1 month
  incidence of bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Shengqing Li, Ph D, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan hospital,Fudan university, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Aleva FE, Voets LWLM, Simons SO, de Mast Q, van der Ven AJAM, Heijdra YF. Prevalence and Localization of Pulmonary Embolism in Unexplained Acute Exacerbations of COPD: A Systematic Review and Meta-analysis. Chest. 2017 Mar;151(3):544-554. doi: 10.1016/j.chest.2016.07.034. Epub 2016 Aug 12. PMID 27522956
- [Background] Wang F, Cheng ZZ, Wang JL, Han WZ, Sun NN. [Incidence of pulmonary embolism in patients with acute exacerbations of chronic obstructive pulmonary disease: a meta-analysis]. Zhonghua Yi Xue Za Zhi. 2013 Jun 25;93(24):1868-71. Chinese. PMID 24124736
- [Background] Akpinar EE, Hosgun D, Akpinar S, Atac GK, Doganay B, Gulhan M. Incidence of pulmonary embolism during COPD exacerbation. J Bras Pneumol. 2014 Jan-Feb;40(1):38-45. doi: 10.1590/S1806-37132014000100006. PMID 24626268
- [Background] Kearon C, Akl EA, Ornelas J, Blaivas A, Jimenez D, Bounameaux H, Huisman M, King CS, Morris TA, Sood N, Stevens SM, Vintch JRE, Wells P, Woller SC, Moores L. Antithrombotic Therapy for VTE Disease: CHEST Guideline and Expert Panel Report. Chest. 2016 Feb;149(2):315-352. doi: 10.1016/j.chest.2015.11.026. Epub 2016 Jan 7. PMID 26867832
- [Background] Chen CY, Liao KM. The Incidence of Deep Vein Thrombosis in Asian Patients With Chronic Obstructive Pulmonary Disease. Medicine (Baltimore). 2015 Nov;94(44):e1741. doi: 10.1097/MD.0000000000001741. PMID 26554770
- [Background] EINSTEIN-PE Investigators; Buller HR, Prins MH, Lensin AW, Decousus H, Jacobson BF, Minar E, Chlumsky J, Verhamme P, Wells P, Agnelli G, Cohen A, Berkowitz SD, Bounameaux H, Davidson BL, Misselwitz F, Gallus AS, Raskob GE, Schellong S, Segers A. Oral rivaroxaban for the treatment of symptomatic pulmonary embolism. N Engl J Med. 2012 Apr 5;366(14):1287-97. doi: 10.1056/NEJMoa1113572. Epub 2012 Mar 26. PMID 22449293
- [Background] Ageno W, Mantovani LG, Haas S, Kreutz R, Haupt V, Schneider J, Turpie AG. XALIA: rationale and design of a non-interventional study of rivaroxaban compared with standard therapy for initial and long-term anticoagulation in deep vein thrombosis. Thromb J. 2014 Jul 14;12:16. doi: 10.1186/1477-9560-12-16. eCollection 2014. PMID 25093014
- [Background] Cohen AT, Spiro TE, Buller HR, Haskell L, Hu D, Hull R, Mebazaa A, Merli G, Schellong S, Spyropoulos AC, Tapson V; MAGELLAN Investigators. Rivaroxaban for thromboprophylaxis in acutely ill medical patients. N Engl J Med. 2013 Feb 7;368(6):513-23. doi: 10.1056/NEJMoa1111096. PMID 23388003
- [Background] Duran A, Sengupta N, Diamantopoulos A, Forster F, Kwong L, Lees M. Cost and outcomes associated with rivaroxaban vs enoxaparin for the prevention of postsurgical venous thromboembolism from a US payer's perspective. J Med Econ. 2011;14(6):824-34. doi: 10.3111/13696998.2011.623203. Epub 2011 Oct 24. PMID 22023098